CLINICAL TRIAL: NCT01266395
Title: Impact of Morning Symptoms in Clinical Control of COPD
Brief Title: Impact of Morning Symptoms in Clinical Control of Chronic Obstructive Pulmonary Disease (COPD)
Acronym: IMPAEPOC
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca
Other Study IDs: NIS-RES-DUM-2010/2
Record Dates: First submitted 2010-12-21; First posted 2010-12-24 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-08

CONDITIONS: COPD
Keywords: morning symptoms COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Observational study to know the Impact of morning symptoms in clinical control of COPD patients. 1200 patients will be included by General practitioners (GPs) and pneumologists. Objective: establish if there are differences in the impact of COPD on daily activities and morning symptoms measured through questionnaires of daily life activity (Capacity of Daily Living during the Morning (CDLM), Global Chest Symptoms Questionnaire (GCSQ))

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed informed consent form
* Patients of both sexes,> 40 years.
* Patients diagnosed with COPD according to global consensus on the definition, classification and management of the disease (GOLD) criteria:

  * post-bronchodilator forced expiratory volume in 1 s (FEV1) / forced vital capacity (FVC) <70%
  * post-bronchodilator FEV1 <80% (stage II, III and IV)

Exclusion Criteria:

* Participating in an epidemiological study or clinical trial
* Patient with other respiratory disease than COPD (eg bronchial asthma, cystic fibrosis, severe bronchiectasis, restrictive lung disease, cancer, etc.).
* Patients with mild COPD: FEV1> 80%

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General Practitioners and pneumologist
Sampling Method: Probability Sample
Enrollment: 1268 (Actual)
Dates: Start 2010-01; Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Determine if there are differences in the impact of COPD on patients according to the characteristics of the disease. To measure the impact of specific self-administered questionnaires used in COPD: CDLMQ, GCSQ and CCQ | Retrospective, (previous 24 months)
  Capacity of Daily Living during the Morning Qustionnaire (CDLMQ), Global Chest Symptoms Questionnaire (GCSQ)and COPD Control Questionnaire (CCQ)

SECONDARY OUTCOMES:
Assess comorbidities as a risk factor for frequent exacerbations | Retrospective, (previous 24 months)

CONTACTS AND LOCATIONS:
Locations (52):
- Spain (52):
  - Research Site, Vitoria-Gasteiz, Alava
  - Research Site, Elda, Alicante
  - Research Site, Petrel, Alicante
  - Research Site, Almería, Almeria
  - Research Site, Ávila, Avila
  - Research Site, Badajoz, Badajoz
  - Research Site, Inca, Balearic Islands
  - Research Site, Son Ferriol, Balearic Islands
  - Research Site, Barcelona, Barcelona
  - Research Site, El Hospitalet de Llobregat, Barcelona
  - Research Site, Puerto Real, CAdiz
  - Research Site, Castellon, Castellon
  - Research Site, Torreblanca, Castellon
  - Research Site, Vinaròs, Castellon
  - Research Site, Lucena, Cordoba
  - Research Site, Pea'arroya-pueblonuevo, Cordoba
  - Research Site, A Picota (mazaricos), Coruna
  - Research Site, Carballo (carballo), Coruna
  - Research Site, Ferrol, Coruna
  - Research Site, Santiago de Compostela, Coruna
  - Research Site, Guadalajara, Guadalajara
  - Research Site, Donostia / San Sebastian, Guipuzcoa
  - Research Site, Placencia de Las Armas-soraluz, Guipuzcoa
  - Research Site, Espelúy, Jaen
  - Research Site, Mures, Jaen
  - Research Site, Nájera, La Rioja
  - Research Site, Arguineguín, Las Palmas
  - Research Site, Abadin (casco Urbano), Lugo
  - Research Site, Baralla (casco Urbano), Lugo
  - Research Site, Lugo, Lugo
  - Research Site, Viveiro (casco Urbano), Lugo
  - Research Site, Alcalá de Henares, Madrid
  - Research Site, Alcorcón, Madrid
  - Research Site, Madrid, Madrid
  - Research Site, San Sebastián de los Reyes, Madrid
  - Research Site, Cieza, Murcia
  - Research Site, Murcia, Murcia
  - Research Site, Pamplona, Navarre
  - Research Site, Leiro (capital), Ourense
  - Research Site, Vigo, Pontevedra
  - Research Site, Arriondas, Principality of Asturias
  - Research Site, Cangas de Narcea, Principality of Asturias
  - Research Site, Jarrio, Principality of Asturias
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, Dos Hermanas, Sevilla
  - Research Site, Seville, Sevilla
  - Research Site, Villanueva del Ariscal, Sevilla
  - Research Site, Benaguasil, Valencia
  - Research Site, Burjassot, Valencia
  - Research Site, La Pobla de Vallbona, Valencia
  - Research Site, Valencia, Valencia
  - Research Site, Zaragoza, Zaragoza